CLINICAL TRIAL: NCT05536895
Title: C-arm Cone Beam CTP Guided Cerebrovascular Interventions: Evaluating Predictability and Accuracy for the Treatment of Acute Cerebral Ischemia in the Angiography Suite
Brief Title: C-arm Cone Beam CTP Guided Cerebrovascular Interventions
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: There is now a commercially available product, the evidence from this study is no longer required to justify adoption of perfusion imaging in the angio suite.
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015-0482 Phase 2; 1U01EB021183-01 (NIH); A539300 (Other: UW Madison); SMPH\RADIOLOGY\RADIOLOGY (Other: UW Madison); Protocol Version 10/13/2021 (Other: UW Madison)
Record Dates: First submitted 2022-09-08; First posted 2022-09-13 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Acute Ischemic Stroke
Keywords: Stroke
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — Multidetector Computed Tomography

STUDY DESIGN:
Intervention Model Description: Single center, randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- C-ARM CBCT (Experimental): A C-arm CBCT evaluation with SMART RECON novel software for the rapid assessment of time-resolved CT angiogram and CT perfusion.
  Interventions: Diagnostic Test: C-Arm Cone Beam Computed Tomography
- MD-CT (Active Comparator): An evaluation with conventional, standard of care, multi-detector CT (MD-CT)
  Interventions: Diagnostic Test: Multi-detector Computed Tomography

INTERVENTIONS:
Diagnostic Test: C-Arm Cone Beam Computed Tomography — C-ARM CBCT angiogram and CBCT perfusion imaging using prototype software (SMART-RECON) can rapidly and accurately assess the cerebral blood flow maps in the setting of decreased blood flow to the brain (ischemic cerebrovascular events). This rapid assessment would eliminate the need for the patient to be imaged in another scanner and be subsequently transported again to another room; all anatomic and physiologic imaging would occur in the angiography suite.
  Other Names: C-ARM CBCT
  Arms: C-ARM CBCT
Diagnostic Test: Multi-detector Computed Tomography — Conventional, standard of care perfusion imaging for AIS
  Other Names: MD-CT
  Arms: MD-CT

SUMMARY:
The study objective for the Phase 2 of this research is to demonstrate and confirm the substantial time savings that can be obtained using cone beam computed tomography (CB-CT) for both complete image acquisition and rapid image reconstruction in a Direct to Angio paradigm (One Stop Shop) for selected acute ischemic stroke (AIS) patients.

DETAILED DESCRIPTION:
Phase 2 of this research is aimed at validating the feasibility and time savings of bringing selected acute ischemic stroke patients with suspected large vessel occlusion directly on hospital arrival to the angiography suite, avoiding the emergency room and conventional MD-CT imaging. In order to make this phase of the study more robust and to reduce bias on image assessment we will prospectively randomize the patients in a 2:1 fashion to either direct to angio for CB-CT imaging or MD-CT imaging in the emergency room. A total of 60 CB-CT subjects and 30 MD-CT subjects will comprise this cohort. Entrance criteria will be identical to those in Phase 1, except the NIHSS must be greater than 8 which is clinically correlative with a likely large vessel occlusion and, since this is standard of care imaging for acute ischemic stroke, GFR will be removed as an exclusionary criteria.

The Phase 1 of this research was registered to NCT03232151.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with acute ischemic stroke presenting within 24 hours of onset
2. Patients that present with a large artery occlusion
3. Adults 18 years of age or older.
4. Patients of childbearing potential must not be pregnant.
5. National Institutes of Health Stroke Scale (NIHSS) of <8
6. No severe co-morbidities

Exclusion Criteria:

1. Patients that are pregnant
2. History of severe renal disease (e.g. stage 4-5)
3. History of renal transplant

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility measured as the amount of time from hospital arrival to the angiography suite | 1 visit (up to 120 minutes)
  Phase 2 of the human subject study aims to further assess the feasibility as a measure the amount of time it takes to bring selected acute ischemic stroke patients with suspected large vessel occlusion directly on hospital arrival to the angiography suite, avoiding the emergency room and conventional MD-CT imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Aagaard-Kienitz, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No